CLINICAL TRIAL: NCT02349776
Title: How do Stories of Survival Help Patients Going Through Bone Marrow Transplant?
Brief Title: Experiencing Transplant With Stories From Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GS12/10259
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients for allograft transplant (Experimental): For the testimonial part all patients who have received an allograft transplant in the last five years will be eligible for participation if they have capacity to consent and can speak English fluently.
  Interventions: Other: Providing testimonies from survivors of transplants to patients

INTERVENTIONS:
Other: Providing testimonies from survivors of transplants to patients — Patients will be asked to complete one mood measure (the HADS), the Life Orientation Test (LOT), and a questionnaire about expectations of treatment in clinic once a decision to proceed to transplant has been made.
  Patients will receive the testimonies upon admittance to the transplant unit and then receive the HADS and a structured interview within the first week of being admitted to the transplant ward (just prior to receiving the transplant) and within the first two weeks following the transplant.

SUMMARY:
Allograft transplants are offered to people with haematological cancers sometimes as the best chance of a cure. However, the survival rates for these procedures can be quite poor, as the transplant, in itself, can be lifethreatening.

In addition, these procedures usually involve a period of lengthy hospitalisation accompanied by a host of debilitating conditions which patients must cope with in isolation due to their increased risk of serious infection. Perhaps unsurprisingly, there is considerable evidence that mood plays a role in the way people recover.

I wish to investigate the psychological impact of providing testimonies from survivors of transplants to patients undergoing the procedure.

The plan is initially to collect about 10-15 testimonials from past transplant patients using a videotaped structured interview then to collate these testimonials into a booklet format and DVD.

This booklet and DVD would be used as an intervention where 40 consecutive patients who are going ahead for transplant are invited to receive the testimonial intervention.

Patients will be asked to complete one mood measure (the HADS), the Life Orientation Test (LOT), and a questionnaire about expectations of treatment in clinic once a decision to proceed to transplant has been made. Patients will receive the testimonies upon admittance to the transplant unit and then receive the HADS and a structured interview within the first week of being admitted to the transplant ward (just prior to receiving the transplant) and within the first two weeks following the transplant.

Comparative analyses of the measures between the three time points would be performed and qualitative analysis of the structured interview data.

Around 80 people undergo transplant each year, it is estimated that the project will be completed by September 2016. The intention would be to publish following completion.

ELIGIBILITY:
Inclusion Criteria:

* For the testimonial part all patients attending bone marrow transplant follow-up clinic who have had an allogenic transplant and who have capacity to consent to the study and who are fluent in English will be eligible.

For the intervention part all patients going forward for allogenic transplant at St James's Institute for Oncology who have capacity to consent to the study and who are fluent in English will be eligible.

Exclusion Criteria:

* Patients without capacity to consent will not be eligible for participation Patients who are not fluent in English will not be eligible for participation Patients who are not going forward for allogenic transplant will not be eligible

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Structured interviews | 3 months
  The short structured interviews investigating patient's experience of the intervention at two time-points following the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom